CLINICAL TRIAL: NCT00492193
Title: A Prospective, Observational, Multi-center Study Assessing Early Post-Operative Recovery Following Laparoscopic Partial Large Bowel Resection
Brief Title: Early Post-Op Recovery After Partial Large Bowel Resection
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Conor Delaney, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 01-07-14; 14CL401 (Other: Adolor Corporation)
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2008-08

CONDITIONS: Diverticulitis; Colon Polyps; Colorectal Cancer
Keywords: Hand assist laparoscopic partial large bowel resection; Laparoscopic partial large bowel resection
MeSH Terms: conditions — Diverticulitis; Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to gather information on the postoperative recovery time and hospital length of stay experienced by patients having laparoscopic surgeries. This trial will also collect data on daily surgical pain and pain medication and how it relates to recovery after surgery. In addition, the investigators will collect data on the use of pain medication and laxatives in patients following laparoscopic large bowel resection.

DETAILED DESCRIPTION:
Laparoscopic surgery was initially performed by surgeons in France in 1987 and was introduced in the United States in 1988. This minimally invasive procedure was performed for cholecystectomy, and is now the standard of care in the treatment of gallbladder disease. Recent advances in laparoscopic surgery and its success in cholecystectomy have permitted the procedure to be used for treating a variety of diseases and for diagnosing and staging.

Minimally invasive laparoscopic surgery has advantages over conventional open surgery, including smaller incisions, earlier gastrointestinal (GI) recovery, shorter hospital stays, less pain, and fewer complications. In recent years evidence is accumulating for some operations that laparoscopic procedures produce outcomes that are comparable to those produced by routine open surgery and may actually surpass others.

Whereas laparoscopic surgery has been successful and well accepted for various abdominal and pelvic surgeries, its use in the area of colorectal surgery has progressed at a slower rate. There are challenges impacting the wider use of laparoscopic bowel resection (LBR). These include the technical difficulty associated with the size of the colon, the need for complete immobilization of the bowel and the need for a watertight, non-leaking anastomosis. In addition, the equipment is expensive and surgeons require specialized training.

Results from studies in colon cancer now indicate that LBR reduces perioperative morbidity, and decreases hospital stay with comparable cancer-related survival as compared to open colectomy. The use of LBR in short-term outcomes is increasing because clinical trial data have demonstrated superiority of LBR, particularly in short-term outcomes over conventional open surgery.

Gastrointestinal recovery and related patient outcomes during the early postoperative period following open segmental colon resection have been extensively evaluated in previous randomized, controlled, multicenter trials. Current data in laparoscopic colectomy have been collected from retrospective, single center clinical trials which lacked standardized definitions and endpoints. Therefore, this prospective, multicenter study in LBR is being undertaken to determine how this surgical technique impacts GI recovery and related outcomes relative to the open laparotomy.

The primary objective of this study is to assess the clinical course of gastrointestinal (GI) recovery and hospital length of stay in subjects undergoing laparoscopic partial large bowel resection. The secondary objective is to assess the immediate post discharge clinical course of subjects undergoing laparoscopic bowel resection with respect to opioid-induced GI effects, daily surgical pain, opioid consumption and laxative use.

ELIGIBILITY:
Inclusion Criteria:

* be male or female at least 18 years of age
* be scheduled for laparoscopic (SL or HAL) partial large bowel resection with primary anastomosis.
* have an American Society of Anesthesiologists Physical Status Score of P1 to P3 (Appendix C.1 of the full protocol).
* are scheduled to receive postoperative pain management primarily with opioid analgesia via intravenous (IV) patient-controlled analgesia (PCA)
* are scheduled to have the NG tube removed on the morning of POD 1
* are able to read, write, and fully understand the language of the study diary
* be able to understand the study procedure, agrees to participate in the study program, and voluntarily provides informed consent.

Exclusion Criteria:

* be scheduled for a total colectomy, ileal pouch-anal anastomosis, colostomy, ileostomy, right HAL colectomy or have a history of total colectomy, gastric bypass, previous bowel resection or short bowel syndrome.
* has a complete bowel obstruction
* has taken therapeutic doses of opioids for 7 consecutive days immediately before surgery.
* has participated in a clinical trial with alvimopan or has taken alvimopan in the past 30 days.
* has a diagnosed history of alcoholism or drug addiction (eg, opioids or other drugs of abuse) within 1 year of the surgery date (Day 0).
* has a diagnosed history of constipation, pelvic floor disorder, or GI disorders known to affect bowel function (eg, chronic diarrhea)
* has a history of laxative dependence or daily use (ie, hyperosmotics, mineral oil, saline, stimulants, bulking agents, suppositories, lubricants, enemas, or any other natural products that promote bowel motility or cleansing)
* has, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, GI, metabolic disorders or mental conditions (e.g., depression, psychosis) that might confound the results of the study or pose additional risk to the subject.
* has participated in another investigational drug or medical device study within the last 30 days or will be enrolled in another investigational drug or medical device study or any study in which active patient participation is required outside normal hospital data collection during the course of this study.
* is unwilling or unable to complete the study diary.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal Surgery clinic population
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to upper and lower GI recovery and post-operative hospital length of stay. | One year
  The primary outcome or end points were time to upper and lower GI recovery (GI-2: tolerance of solid food and bowel movement) and post-operative hospital length of stay.

SECONDARY OUTCOMES:
Postoperative ileus related mobidity. | One year
  The secondary outcome or endpoints are postoperative ileus(POI) related morbidity (postoperative nasogastric tub insertion or investigator-assisted POI resulting in prolonged hospital stay or readmission), conversion rate, and protocol-defined prolonged POI (GI-2>5 postoperative days.)

CONTACTS AND LOCATIONS:
Overall Officials: Conor P. Delaney, MD, PhD, Principal Investigator — University Hospitals of Cleveland/ Institute for Surgical Innovation
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Delaney CP, Marcello PW, Sonoda T, Wise P, Bauer J, Techner L. Gastrointestinal recovery after laparoscopic colectomy: results of a prospective, observational, multicenter study. Surg Endosc. 2010 Mar;24(3):653-61. doi: 10.1007/s00464-009-0652-7. Epub 2009 Aug 18. PMID 19688390